CLINICAL TRIAL: NCT07111013
Title: A 12-Month, Multicenter, Open-Label Extension (OLE) Study to Assess the Long-Term Safety of Lifitegrast/Perfluorohexyloctane Fixed-Dose Combination in Subjects With Dry Eye Disease
Brief Title: A Study to Assess the Long-Term Safety of Lifitegrast/Perfluorohexyloctane Fixed-Dose Combination in Subjects With Dry Eye Disease
Acronym: NGL-Long Term
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Business Decision
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BL-RX01-NGL-1301-LTS
Record Dates: First submitted 2025-08-06; First posted 2025-08-08 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes | interventions — lifitegrast; perfluorohexyl-octan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Lifitegrast/perfluorohexyloctane (PFHO) fixed-dose combination (FDC) (5%/95%) (Experimental): Lifitegrast/perfluorohexyloctane (PFHO) fixed-dose combination (FDC) (5%/95%) packaged in multidose bottles, with 1 topical ocular drop instilled in both eyes (OU) twice daily (BID)
  Interventions: Drug: Lifitegrast/perfluorohexyloctane (PFHO)

INTERVENTIONS:
Drug: Lifitegrast/perfluorohexyloctane (PFHO) — fixed-dose combination (FDC) (5%/95%)

SUMMARY:
A Study to Assess the Long-Term Safety of Lifitegrast/Perfluorohexyloctane Fixed-Dose Combination in Subjects With Dry Eye Disease

ELIGIBILITY:
Inclusion Criteria:

This study will include subjects who meet all of the following inclusion criteria:

1. Voluntarily provide written informed consent
2. Completed Study BL-RX01-OPUSNG-1201 and:

   1. Were compliant with BL-RX01-OPUSNG-1201 trial procedures and study drug use
   2. Had no important protocol deviations
   3. Had no ongoing adverse events (AEs)
3. Are able and willing to follow instructions, including participation in all trial assessments and visits

Exclusion Criteria:

This study will exclude subjects who meet any of the following exclusion criteria (Note: Ocular exclusion criteria are relevant to both eyes, such that meeting a criterion in either eye excludes the subject from the study):

1. Have best-corrected visual acuity (BCVA) of 0.7 logMAR or worse (50 Early Treatment Diabetic Retinopathy Study [ETDRS] letters; Snellen equivalent score of 20/100 or worse) at Visit 1 (Screening/Baseline)
2. Have any clinically significant (CS) ocular surface slit-lamp findings and/or in the opinion of the Investigator have any findings that may interfere with trial parameters
3. Any concurrent condition, concomitant treatment, or situation which, in the Investigator's opinion, may put the subject at significant risk, confound study results, or interfere with their participation in the trial
4. Planned contact lens use during the trial
5. Planned ocular and/or lid surgeries during the trial
6. Unable or unwilling to avoid all topical dry eye treatments (except for study drug) during the first 4 weeks of participation
7. Any non-drug therapies affecting meibomian glands such as LipiFlow® and Intense Pulse Light during the trial
8. Participation in any investigational drug or device study other than BL RX01-OPUSNG-1201 or BL-RX01-NGL-1301-LTS
9. Any female who is nursing, lactating, pregnant, planning a pregnancy, or has a positive urine pregnancy test at Visit 1 (Screening/Baseline)
10. Any female of childbearing potential (FOCBP) who is unwilling to agree to:

    1. Have a urine pregnancy testing performed at Visit 1 (Screening/Baseline)
    2. Use at least 1 medically acceptable form of birth control for at least 14 days prior to the first dose of study drug, throughout the study duration, and for 1 month after the last dose of study drug Note: FOCBPs include all females who have experienced menarche and have not experienced menopause (as defined by amenorrhea for greater than 12 consecutive months) or have not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy)

    Note: Acceptable forms of birth control include:
    * Mechanical (spermicide in conjunction with a barrier such as a diaphragm or condom)
    * Hormonal contraceptive (oral, injectable, implantable, or transdermal)
    * Intrauterine device
    * Surgical sterilization of male partner at least 3 months prior to the first dose of study drug Note: For non-sexually active female subjects, abstinence may be regarded as an adequate method of birth control when this is in line with the preferred and usual lifestyle of the subject; however, if the subject becomes sexually active during the trial, she must agree to use adequate birth control as defined above for the remainder of the trial
11. Any male who is unwilling to agree to use at least 1 medically acceptable form of birth control with female partner (FOCBP)

Note: Acceptable forms of birth control include:

* True abstinence (when this is in line with the preferred and usual lifestyle of the subject), or
* Vasectomy at least 3 months prior to the first dose of study drug Without a vasectomy, must use condoms with spermicidal foam, gel, film, cream, suppository at least 14 days prior to the first dose of study drug, throughout the study duration, and for 1 month after the last dose of the study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment Emergent Adverse Events | Assessed for 12 months